CLINICAL TRIAL: NCT02299297
Title: An Open-Label Pilot Study To Evaluate The Efficacy Of Tofacitinib In Moderate To Severe Alopecia Areata, Totalis And Universalis
Brief Title: Study To Evaluate The Efficacy Of Tofacitinib In Moderate To Severe Alopecia Areata, Totalis And Universalis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Locks of Love (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO1502
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tofacitinib (Experimental): Tofacitinib will be self-administered for 6 months, with the option to extend treatment up to an additional 6 months at the discretion of the principal investigator. Patients will then be followed for 6 months off the drug to assess the incidence and timing of recurrence of disease or documentation of delayed response to treatment.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Dosage/Frequency: 5mg - 10mg, oral, twice daily
  Other Names: XELJANZ

SUMMARY:
This is an open-label pilot study of tofacitinib taken daily for 6 months in the treatment of moderate to severe AA, and alopecia totalis or universalis, followed by 6 months follow-up off drug to assess the incidence and timing of recurrence of disease or documentation of delayed response to treatment. There will be the option of increasing the treatment duration up to an additional 6 months beyond the initially scheduled 6 months of treatment, if clinically indicated, and at the discretion of the investigator.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a common disease of the immune system, known as an "autoimmune" disease. In the disease, the immune system mistakenly destroys the hair follicle, causing hair to fall out. Despite many people having this disease, research into its cause and new, better ways to treat AA has lagged far behind other similar diseases of the immune system. Currently, there are no Federal Drug Administration approved drugs for AA.

Tofacitinib (made by Pfizer) is an intervention known to effectively treat a disease of the joints, known as rheumatoid arthritis. It is also being studied in the treatment of psoriasis, another "autoimmune" disease, by fighting inflammation. There are some genetic and chemical similarities between those with active rheumatoid arthritis, psoriasis, and AA,suggesting that treatment with the same drug is likely to be effective. In mice specially designed for testing drugs for the treatment of human alopecia, this medication worked to prevent the disease AA from starting in mice that would have otherwise developed the disease. To test Tofacitinib, we are going to treat 15 patients with moderate to severe AA for up to 6 months. This is an "open label" study, meaning that there will not be a placebo group; all patients enrolled in the study will receive the active medication. The effectiveness of the medication will be measured by changes in hair re-growth as determined by physical exam and photography, as well as by patient and physician scoring. After the treatment period of up to 6 months is completed, There will be the option of increasing the treatment duration up to an additional 6 months beyond the initially scheduled 6 months of treatment, if clinically indicated, and at the discretion of the investigator. Patients will be followed for another 6 months off of the drug to see if the effects of treatment last and if there is delayed response. The safety of the medication, Tofacitinib, in patients with AA will also be evaluated. Blood work will be collected before medication is started, during the treatment period and after Tofacitinib is stopped in order to monitor for adverse effects of the medication. Small scalp biopsies and peripheral blood will be taken at the beginning of the study before treatment and at weeks 4 and 24. Additional, optional scalp biopsies and blood draws may be suggested at other important time points. The chemical analysis of these skin samples and blood will help us to understand how the disease happens, how the treatment works, and even guide us to better treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age.
* Patients with a diagnosis of moderate to severe patch type alopecia areata.
* Patients with alopecia totalis or universalis may be enrolled.
* Patients have >30% and <95% total scalp hair loss at baseline as measured using the SALT score to qualify as moderate to severe patch type AA; and 95-100% scalp hair loss to qualify as alopecia totalis or universalis.
* Duration of hair loss greater than 3 months without an upper limit of duration as long as there is reason to believe that regrowth is possible in the opinion of the investigator.
* No evidence of significant active ongoing regrowth present at baseline.
* Patients with a history of alopecia totalis/universalis can be included as long as the current episode of hair loss meets the criteria of 30 to 95% hair loss (i.e. they are not currently AT or AU), and as long as in the opinion of the investigator there does appear to be potential for regrowth. Patients with current episodes of alopecia totalis/universalis may be included in this study.
* Vaccinations should be up to date in agreement with current immunization guidelines prior to start of tofacitinib. The patient will be asked to obtain verbal verification from their primary care provider that this is the case.
* Patients may be naïve to treatment or unresponsive to intralesional (IL) steroids or other treatments for alopecia areata.
* Women of childbearing potential (WOCBP) must use highly effective methods of birth control [for at least 12 weeks after the last dose of investigational product] to minimize the risk of pregnancy. WOCBP must follow instructions for birth control for the entire duration of the study including a minimum of 90 days after dosing has been completed.

Acceptable methods of highly effective birth control include:

* Condom with spermicide
* Diaphragm and spermicide
* Cervical cap and spermicide The use of intrauterine devices, (IUDs) shall be at the discretion of the investigator.

  1. Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
  2. Women must not be breastfeeding.

Exclusion Criteria:

* Sex and Reproductive Status

  1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 12 weeks after the last dose of study drug.
  2. WOCBP using a prohibited contraceptive method.
  3. Women who are pregnant or breastfeeding.
  4. Women with a positive pregnancy test on enrollment or before administration of tofacitinib.
  5. Sexually active fertile men not using effective birth control if their partners are WOCBP.
* Target Disease Exceptions

  1. Patients with current alopecia totalis/universalis (i.e. 100% scalp or 100% scalp and body loss, respectively) may be enrolled.
  2. Patients with a history of or active skin disease on the scalp such as psoriasis or seborrheic dermatitis.
  3. Patients in whom the diagnosis of alopecia areata is in question or in whom the pattern of hair loss is such that quantification of hair loss and assessment of regrowth is difficult. E.g patients with diffuse alopecia areata. This assessment is at the investigator's discretion.
  4. Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma) that in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections.
  5. Patients with hemoglobin levels <9 g/dL, lymphocyte count <500 cells/mm3, absolute neutrophil count (ANC) <1000 cells/mm3, at baseline.
  6. Patients known to be HIV or hepatitis B or C positive.
  7. Patients with history or evidence of moderate or severe hepatic and/or renal impairment.
  8. Patients with history of immunosuppression or history of recurrent serious infections.
* Coexisting disease or concurrent medications

  1. Patients taking potent inhibitors of CYP3A4 (e.g.ketoconazole).
  2. Patients receiving one or more concomitant medications that result in both moderate inhibition of CYP3A4 and potent inhibition of CYP2C19 (e.g., fluconazole).
  3. Patients known to be HIV or hepatitis B or C positive.
  4. Patients with evidence of infection or active/untreated skin cancer.
  5. Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, diphenylcyclopropenone (DPCP), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth within one month of the baseline visit.
  6. Patients who are impaired, incapacitated, or incapable of completing study-related assessments.
  7. Patients with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
  8. Female patients who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
  9. Patients with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ. Existing non-melanoma skin cell cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug.
  10. Patients who currently abuse drugs or alcohol.
  11. Patients with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
  12. Patients with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
  13. Patients who have received any live vaccines within 3 months of the anticipated first dose of study medication. Subjects may not receive live vaccine concurrently with tofacitinib.
  14. Patients with a history or symptoms suggestive of gastrointestinal perforation or disorders that might increase the risk of GI perforation such as gastric ulcers or diverticulitis.
  15. Patients who take NSAIDs at high dose or on a frequent basis, which in the investigator's opinion might increase the risks of gastrointestinal perforation.
  16. Patients with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (e.g., chronic pyelonephritis, osteomyelitis, or bronchiectasis).
  17. Patients at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (4 weeks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be included in the publications, but will not be identifiable.
Time Frame: At the end of the study.
Access Criteria: The data is available in the publication for this study.

REFERENCES:
- [Derived] Jabbari A, Sansaricq F, Cerise J, Chen JC, Bitterman A, Ulerio G, Borbon J, Clynes R, Christiano AM, Mackay-Wiggan J. An Open-Label Pilot Study to Evaluate the Efficacy of Tofacitinib in Moderate to Severe Patch-Type Alopecia Areata, Totalis, and Universalis. J Invest Dermatol. 2018 Jul;138(7):1539-1545. doi: 10.1016/j.jid.2018.01.032. Epub 2018 Feb 13. PMID 29452121

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tofacitinib
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Includes all individuals who received treatment.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Responders
Description: This is defined as 50% or greater hair re-growth from baseline as assessed by the Severity of ALopecia Tool (SALT) score after up to 24 weeks/6 months to 72 weeks/18 months of treatment. This is a relatively strict definition for defining responders and non-responders and was chosen to minimize the potential for spontaneous remission, in which fewer than 10% are expected to achieve this magnitude of hair regrowth spontaneously.
Time Frame: Baseline up to between 24 and 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 12
Participants | 8

2. Secondary Outcome: Total Number of Responders Maintaining Response During the Post-Treatment Follow Up Period
Description: To assess the durability of responses, patients who achieve 50% regrowth from baseline during the first 6 to 18 months, will continue to be followed for an additional 6 months post-treatment or until it is determined that relapse has occurred. Durability of response was measured by comparing SALT scores from baseline to 24 weeks after treatment.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 8
Participants | 3

3. Secondary Outcome: Total Number of Responders With Change in PHYSICIAN Global Assessment Score
Description: A physician's assessment of the severity of disease based on a 6-point scale (score of 0 = clear and 5 = very severe). Responders are defined by participants who exhibited regrowth.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 8
Participants | 8

4. Secondary Outcome: Percentage of Regrowth
Description: Percentage of regrowth was measured by comparing the SALT score at the beginning and end of treatment.
Time Frame: Baseline up to between 24 and 72 weeks
Measure: Mean (Full Range); unit: percentage of regrowth
Arm/Group | Tofacitinib
Number analyzed (Participants) | 12
percentage of regrowth | 56.8 [12.1 to 100]

5. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: The first dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire used to evaluate patient's quality of life. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 12
score on a scale
  Baseline | 6.5 (5.0)
  3 months | 5.2 (6.7)
  6 months | 6 (6.9)

ADVERSE EVENTS:
Time Frame: Up to 18 months from the start of treatment
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib (N=12)
Upper respiratory infection (Infections and infestations) | 11 (11)
increased bowel movement frequency (Renal and urinary disorders) | 4 (4)
Blood on urinalysis (Blood and lymphatic system disorders) | 4 (4)
Loose stools (Metabolism and nutrition disorders) | 3 (3)
Mild acne (General disorders) | 3 (3)
Weight gain (Metabolism and nutrition disorders) | 2 (2)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2)
Hypertensive urgency (Vascular disorders) | 1 (1)
Bloating (General disorders) | 1 (1)
Constipation (Metabolism and nutrition disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Neuropathic pain (Nervous system disorders) | 1 (1)
Vaginal spotting (post menopause) (Reproductive system and breast disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT02299297/Prot_SAP_000.pdf